CLINICAL TRIAL: NCT06225544
Title: Lumasiran in Hyperoxalaemic Patients on Haemodialysis
Acronym: LHOxH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Alnylam Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Gerlineke Hawkins-van der Cingel, Deputy PI, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20018510; 2022-002681-32 (EudraCT Number)
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Haemodialysis; Chronic Kidney Disease Requiring Chronic Dialysis; Cardiovascular Disease; Cardiovascular Risk Factor; Hyperoxalemia
MeSH Terms: conditions — Cardiovascular Diseases | interventions — lumasiran; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a randomised controlled trial with parallel arms of placebo versus study drug (lumasiran). With a 1:1 ratio between the two groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lumasiran, treatment arm (Experimental): Treatment arm with Lumasiran
  Interventions: Drug: Lumasiran
- Placebo (Placebo Comparator): Placebo injection with 0.9% sodium chloride
  Interventions: Drug: 0.9% Sodium Chloride (placebo)

INTERVENTIONS:
Drug: Lumasiran — Subcutaneous injection, given as three monthly loading doses followed by one further maintenance dose.
  Arms: Lumasiran, treatment arm
Drug: 0.9% Sodium Chloride (placebo) — Placebo, subcutaneous injection, given as three monthly loading doses followed by one further maintenance dose.
  Arms: Placebo

SUMMARY:
This study will look at how well a drug that reduced the amount of oxalate in the body works in patients that have kidney disease and need dialysis treatment. People with kidney disease often have higher levels of oxalate in the blood. People with kidney disease are also at higher risk of having heart attacks, heart disease and strokes (these are called cardiovascular diseases). It is thought that high oxalate levels may increase the risk of these diseases. This study will investigate if this medicine can lower the amount of oxalate in the blood of dialysis patients and see if there is any change in the health of their heart. This medicine is already used for people who have high oxalate levels because of a genetic cause and has been used safely for patients on dialysis.

The study will put the participants randomly into either the group getting the study medicine or the group getting a placebo (this will be a solution of saline water). Neither participants not the doctors will know whether the drug or placebo is given until after the end of the study.

At the start of the study all the participants will have an echocardiogram (an ultrasound of the heart) and again 6 months later at the end of the study. We will also take blood tests once a month when the participants come for dialysis.

DETAILED DESCRIPTION:
This is an investigator-initiated, double-blind, phase II two-centre medications study with an intervention and placebo arm.

The principal objective of this study is to establish if the administration of lumasiran versus placebo can effectively lower pre-dialysis oxalate levels in hyperoxalaemic haemodialysis patients with any cause of ESKD (end stage kidney disease) except known primary hyperoxaluria.

The hypothesis is that compared to placebo, the administration of lumasiran (the study drug) will reduce serum oxalate levels at 3-6 months post first dose in hyperoxalaemic haemodialysis patients.

This study will evaluate the use of lumasiran in haemodialysis patients. Lumasiran will be dosed as per the SmPC published by the European Medicines Agency. Monthly pre-dialysis plasma oxalate measurements will be taken to assess the effect of lumasiran on lowering the oxalate levels versus a placebo. Thus far studies have shown lumasiran to be well tolerated. The tolerability in this patient cohort will be evaluated and monitor inflammatory and cardiovascular biomarkers in addition to cardiac imaging with echocardiograms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Aged between 18 and 80 years old at the start of the study.
* Women of child-bearing potential to consent to either abstinence or the use of contraception during the study period
* Patients must have capacity to give written, informed consent to participate in the study prior to commencing the study. They must be fully aware of the aims, nature, planned interventions and potential risks of participating in the study. This consent must be obtained by the time of participant inclusion.
* Established and stable on haemodialysis for at least 2 months
* Thrice weekly haemodialysis
* In possession of permanent dialysis access - either arterio-venous fistula (AVF) or graft (AVG) or permanent dialysis catheter/tunnelled haemodialysis line (THL).
* ESKD not caused by previously diagnosed primary hyperoxaluria.
* Mean baseline serum oxalate level of ≥20 μmol/L
* No recent (within last 2 months) significant changes to regular medications or diet

Exclusion Criteria:

* Known diagnosis of PH1, 2 or 3; or a pathological mutation documented to cause primary hyperoxaluria.
* Established on haemodialysis for less than 2 months.
* On peritoneal dialysis.
* Combined haemodialysis and peritoneal dialysis.
* Temporary or poorly functioning haemodialysis access
* Pregnancy, planning pregnancy or currently breast feeding.
* Co-morbidity of an enteric disorder such as Inflammatory Bowel Disease (IBD), short gut syndrome, or a malabsorptive disorder.
* Decompensated Liver failure.
* Intercurrent active infection and/or antibiotic treatment.
* Currently on Vitamin C treatment with a daily dose of more than 250mg.
* Terminal illness and/or life expectancy of less than 1 year.
* Currently relapsed or uncontrolled and symptomatic psychiatric disorder preventing compliance with the study.
* Participants institutionalised by court or government order.
* Patients who could be coerced due to dependency on the sponsor, the investigator, the trial sites or test centres.
* Deranged liver function tests: If alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is more than twice the upper limit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-14 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Pre-dialysis Plasma Oxalate concentration | It will be measured at baseline and month 1-6 (weeks 4, 8, 12, 16, 20 and 24).
  The primary endpoint is the percentage change in pre-dialysis plasma oxalate levels in non-primary hyperoxaluria patients with raised plasma oxalate levels who are receiving maintenance haemodialysis.

SECONDARY OUTCOMES:
Absolute change in pre-dialysis mean plasma | Baseline to month 3-6,
  Absolute change in pre-dialysis mean plasma oxalate levels from baseline to month 3-6, comparing the treatment group with the placebo group.
Side effects (tolerability) | Monthly - month 0-6
  Tolerability will be assessed using an adapted FACIT Instrument validated questionnaire (severity of side effects rated on scale between 0 and 4). Again, the answers of the two study arms will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Felix Knauf, MD, Principal Investigator — Charite Universitätsmedizin
Locations (1):
- Charite Universtiätsmedizin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No